CLINICAL TRIAL: NCT01724489
Title: Skeletal Physiology Dysregulation in Obesity: The Role of Growth Hormone
Brief Title: Study of Growth Hormone and Bone in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Pfizer (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2012P002276
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Osteopenia
MeSH Terms: conditions — Obesity; Bone Diseases, Metabolic | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone (Active Comparator): Growth Hormone is Genotropin, provided by Pfizer Inc. It is self administered daily for 18 months using a 5 mg injection pen device. Dose will be titrated based on IGF-1 levels.
  Interventions: Drug: Growth hormone
- Placebo (Placebo Comparator): Placebo will be provided by Pfizer Inc. It will appear identical to active growth hormone and will be administered in the same manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth hormone
  Other Names: Genotropin (Pfizer Inc.)
  Arms: Growth Hormone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Obesity is an important risk factor for osteoporosis and fractures. With the growing prevalence of obesity in the U.S., understanding the pathophysiology of bone loss in this population is of importance to public health. Growth hormone (GH) is a critical mediator of bone homeostasis and is markedly reduced in obesity. Our preliminary data suggest an important role for the GH/insulin-like growth factor 1 (IGF-1) system in the pathogenesis of bone loss in obesity. The development of novel imaging techniques provides an opportunity to investigate the effects of GH on skeletal structure and strength, which will provide insights into the pathogenesis of obesity related bone loss. Understanding the pathophysiology of bone loss in obesity may help identify new treatment targets for this important complication. The investigator hypothesizes that low-dose GH administration for 18 months will improve skeletal health.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 and generally healthy
* BMI ≥ 25 kg/m2
* Bone mineral density (BMD) T score ≤ -1.0 and > -2.5 (as measured by DXA)

Exclusion Criteria:

* For women: amenorrhea for 3 months, pregnancy or breastfeeding, polycystic ovary syndrome
* History of diabetes mellitus, cancer or other serious chronic disease
* Use of osteoporosis medications
* Anemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-08; Primary Completion 2018-11-15 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miller, MD, Principal Investigator — Massachusetts General Hospital; Miriam Bredella, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from August 2013 to April 2017. Recruitment techniques included posting advertisements on the internet (i.e. Facebook and Craigslist) and on the Massachusetts General Hospital's clinical trial recruitment website.
Pre-assignment Details: Of the 253 people who signed a consent form, 165 were unable to participate due to various reasons including meeting ineligibility criteria. The 88 subjects remaining were randomized to one of two arms. Of these 88 subjects, a total of 77 subjects had baseline measurements collected.
Groups:
- Growth Hormone: Growth Hormone (GH) is Genotropin, provided by Pfizer Inc. It is a self-administered sub-cutaneous daily injection using an injection pen device. It was administered up to 18 months. The dose was titrated based on IGF-1 hormone levels with the goal of maintaining an IGF-1 level in the upper-quartile of the normal range.
- Placebo: Placebo was provided by Pfizer Inc. It appeared identical to active growth hormone and was administered in the same manner; self administered sub-cutaneous daily for 18 months using an injection pen device. Dose was titrated in a way to maintain the double-blind.
Period: Overall Study
Arm/Group | Growth Hormone | Placebo
Started | 39 | 38
Completed | 23 | 26
Not Completed | 16 | 12
Not completed — Adverse Event | 8 | 3
Not completed — Surgery, medication | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Growth Hormone: Growth Hormone is Genotropin, provided by Pfizer Inc. It is self administered daily for 18 months using a 5 mg injection pen device. Dose will be titrated based on IGF-1 levels.
  Growth hormone
- Placebo: Placebo will be provided by Pfizer Inc. It will appear identical to active growth hormone and will be administered in the same manner.
  Placebo
- Total: Total of all reporting groups
Arm/Group | Growth Hormone | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 49 (12) | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 37 | 34 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 27 | 30 | 57
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: Change in BMD over 18 months in the GH vs placebo group
Time Frame: baseline and 18 months
Population: Two subjects from the growth hormone arm were not analyzed due to large amount of weight loss, which has a well-documented effect of decreasing BMD. AP spine bone density in one study subject in the placebo group was excluded because the scan was technically poor.
  These data were excluded before the study was unblinded.
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Growth Hormone | Placebo
Number analyzed (Participants) | 21 | 25
grams/cm^2 | -0.015 (0.033) | -0.008 (0.034)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Growth hormone (Pfizer) is FDA approved and has a possible side-effect profile described/listed in the medication package insert. The investigators recorded all adverse events (as defined by the clinicaltrials.gov definition) and categorized them by "expected" (eg listed in the medication package insert) and "unexpected" (not listed in the medication package insert).
  # of events = # of subjects that experienced the side effect at any point during the study.
Arm/Group | Growth Hormone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/38
Other Adverse Events (participants affected / at risk) | 29/39 | 13/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=39) | Placebo (N=38)
prolonged inpatient psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=39) | Placebo (N=38)
headache (General disorders) | 1 (1) | 2 (3)
edema (swelling) in the hands and/or feet (Blood and lymphatic system disorders) | 8 (11) | 6 (6)
pain and/or stiffness in the hands and/or feet (Musculoskeletal and connective tissue disorders) | 9 (10) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
tingling (Nervous system disorders) | 13 (16) | 3 (4)
myalgia (muscle aches) (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
elevated blood sugar (Metabolism and nutrition disorders) | 5 (5) | 2 (2) — elevated fasting glucose or HbA1c
injection site discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
injection site bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
joint stiffness (not in the hands and/or feet) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study medication was discontinued at 18 months. Subjects were followed for an additional 6 months off of study medication. The data reported here are for the primary 18-month trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT01724489/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT01724489/SAP_001.pdf